CLINICAL TRIAL: NCT05519436
Title: Investigation of the Relationship Between Plantar Foot Pressure and Balance in Morbidly Obese Individuals: A Retrospective Study
Brief Title: Investigation of the Relationship Between Plantar Foot Pressure and Balance in Morbidly Obese Individuals
Status: Completed | Type: Observational
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Gulfidan Tokgoz, Lecturer, Department of therapy and rehabilitation, PhD student, Istanbul University - Cerrahpasa
Other Study IDs: 2022/242
Record Dates: First submitted 2022-08-25; First posted 2022-08-29 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Obesity, Morbid; Foot Deformities
Keywords: plantar pressure; dynamic balance; morbid obesiy; gait
MeSH Terms: conditions — Obesity, Morbid; Foot Deformities | interventions — Restraint, Physical

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Morbid obesity individuals
  Interventions: Other: Assessment
- Healthy individuals
  Interventions: Other: Assessment

INTERVENTIONS:
Other: Assessment — Bioelectrical impedance analysis method was used to evaluate the body composition of the cases. Muscle, fat, water ratio was made with Inbody Bioelectrical Impedance Device. Static and dynamic plantar pressure analyzes were evaluated with Sensor Medica pedobarographic measuring device, and postural sway was evaluated with "bilateral comparison tests", one of the dynamic balance tests of Biodex Balance System.

SUMMARY:
The fact that changes in plantar pressure during walking and in a fixed position in morbidly obese individuals and the relationship between postural oscillations and balance have not been fully elucidated creates a need in this area.

In this study, primary aim is to investigate the change in plantar foot pressure, balance parameters and the relationship between them in morbidly obese individuals compared to healthy individuals.

ELIGIBILITY:
Inclusion Criteria:

* Individuals between the ages of 18-60
* BMI ≥ 40 kg/m2, morbidly obese individual
* No surgical operation in the last 6 months
* Non-obese healthy adult individuals will be included in the study as the control group.

Exclusion Criteria:

* Having a musculoskeletal disorder or systemic disease that will interfere with physical activity
* Presence of balance problems that will prevent physical activity
* Presence of psychiatric or neurological disease affecting cooperation and cognitive functions
* Presence of acute pain
* Presence of uncontrolled diabetes and hypertension
* Having any communication problems

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Morbid obesity (grade 3 or severe obesity), a type of obesity, is defined as BMI equal to or more than 40 kg/m2, and chronic diseases such as increased mortality, diabetes mellitus, hypertension, sleep apnea, cardiovascular, kidney, and lung diseases. It is associated with increased risk of musculoskeletal system diseases and dyslipidemia (3,4).
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
Static and dynamic plantar pressure analyzes | 2019-2020
  To evaluate the plantar pressure, a computerized pedobarographic measuring device with a pressure sensor platform, which can measure the load on the sole of the foot statically and dynamically, and detect the displacement of the pressure center while standing, was used.

SECONDARY OUTCOMES:
Bioelectrical Impedance Analysis (BIA) Measurement | 2019-2020
  The muscle, fat, and water ratio of the cases were evaluated with the Inbody Bioelectrical Impedance Device.
Biodex Balance System | 2019-2020
  Biodex Balance System is a system that provides the opportunity to evaluate the balance statically and dynamically. It allows to measure the displacements in the center of gravity of the patient standing on a standing balance platform and the reactions when the support surface changes. "Bilateral comparison tests", one of the dynamic balance tests of the Biodex balance System, were used to evaluate the postural sway of the cases.

CONTACTS AND LOCATIONS:
Overall Officials: Gulfıdan Tokgoz, Principal Investigator — Istanbul University - Cerrahpasa; Nilay Arman, Principal Investigator — Istanbul University - Cerrahpasa; Ayşenur Namlı, Principal Investigator — Istanbul University - Cerrahpasa; Hakan Seyit, Principal Investigator — BAKIRKOY DR. SADİ KONUK EDUCATION AND RESEARCH HOSPITAL; Mehmet Karabulut, Principal Investigator — BAKIRKOY DR. SADİ KONUK EDUCATION AND RESEARCH HOSPITAL
Locations (1):
- Istanbul University-Cerrahpaşa, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Background] Elrazek AE, Elbanna AE, Bilasy SE. Medical management of patients after bariatric surgery: Principles and guidelines. World J Gastrointest Surg. 2014 Nov 27;6(11):220-8. doi: 10.4240/wjgs.v6.i11.220. PMID 25429323